CLINICAL TRIAL: NCT04225572
Title: Physical Rehabilitation Evaluation and Optimal Physical Therapy (PRE-OPT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2017NTLS119; PMR-2017-26231 (Other: University of Minnesota Masonic Cancer Center)
Record Dates: First submitted 2019-09-24; First posted 2020-01-13 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Patient will not receive physical therapy treatment or further instruction from the research team. The patient will receive standard care recommended by their medical provider which may or may not include physical therapy treatment.
- Physical Therapy Group (Experimental)
  Interventions: Behavioral: Physical Therapy: Dependent on Patient's Needs

INTERVENTIONS:
Behavioral: Physical Therapy: Dependent on Patient's Needs — Therapeutic exercise:
  * ROM: Begin with passive upper extremity ROM and progress to active ROM.
  * Strengthening: Progressive upper extremity resistive exercises starting with light weights.
  * Aerobic: Select a suitable, individual aerobic exercise program (walking, yoga, etc.) Manual therapy
  * Soft tissue mobilization, myofascial release, and stretching of identified tight and stiff tissue.
  Lymphedema treatment
  * Manual lymph drainage: Gentle lymphatic massage to lymph nodes and vessels by PT for 1-2 weeks. Instruct patient in self MLD to perform 1-2×/day for 10 minutes during the remaining weeks.
  * Compression therapy: Gradient compression bandaging for daily wear with activities and exercise for 1-2 weeks. Instruct in self compression bandaging or issue a compression garment to wear with exercise or activity, or with worsening symptoms of AWS (i.e. cording extends down arm) or lymphedema.
  Arms: Physical Therapy Group

SUMMARY:
Phase 1: The investigators will conduct a prospective study to quantify the association between axillary web syndrome (AWS) and metastatic disease and chronic morbidities such as lymphedema, shoulder dysfunction, and pain comparing women (i) with AWS and (ii) without AWS in two cohorts of women. (n=200) Phase 2: This is a randomized controlled trial to 1) quantify the effects of (i) physical therapy compared to (ii) a control group in individuals with AWS following breast cancer surgery related to physical activity and physical impairments such as lymphedema, shoulder motion, function, and pain (n=44, 22 in each group). Funding to progress to Phase 2 of this trial has been obtained. It is anticipated 120 subjects participating in Phase 1 will be screened for eligibility for Phase 2 (separate consent and eligibility from Phase 1).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Patients (female or male) with a tissue diagnosis of non-invasive or invasive breast cancer
* Planned surgical breast cancer treatment (lumpectomy or mastectomy) with a minimum removal of one axillary lymph node by sentinel node biopsy. Contralateral prophylactic mastectomy or bilateral mastectomy is allowed.
* Voluntary written consent signed before performance of any study-related procedure not part of normal medical care

Exclusion Criteria:

* Patients (patients unable to travel easily to the University of Minnesota Medical Center for post-surgery visits).
* Synchronous bilateral breast cancer
* Presence of a medical complication that would prevent the patient from being able to participate in the study, such as terminal cancer
* Previous history of upper extremity deep vein thrombosis
* Breast cancer surgery without lymph node removal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2017-12-27 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2025-12-12 (Actual)

PRIMARY OUTCOMES:
Clinical characteristics of preoperative Auxillary Web Syndrome (AWS) | 1 Year
  Status of lymph nodes in women who have preoperative AWS (lymph node metastasis present or not)
Treatment Effects | 1 Year
  Range of motion (ROM) will be measured using a standard goniometer

SECONDARY OUTCOMES:
Pain level | 1 Year
  Measured by 0-10 scale and Penn Shoulder Score questionaire
Function | 1 Year
  Disabilities of the Arm, Shoulder and Hand questionaire
Lymphedema | 1 Year
  Measured by girth measures, tissue dielectic constant and bioimpedance spectroscopy
Physical activity | 1 Year
  Measured by International Physical Activity Questionaire IPAQ (short form)
Axillary web syndrome status | 1 Year
  (present/not present) based on palpable assessment by investigator
Preoperative AWS and a positive lymph node status | 1 Year
  Correlation between AWS and a positive lymph node status
Abduction range of motion (ROM) | 1 month
  ROM measured by a standard goniometer
DASH Score | 1 Month
  Measured by Disabilities of the Arm, Shoulder, and Hand questionnaire
Body mass index (BMI) | 1 month
  Difference in body mass index (BMI) between patients with and without AWS (pre and post operative)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Koehler, PhD, PT, CLT-LANA, Principal Investigator — University of Minnesota, Division of Physical Therapy
Locations (1):
- University of Minnesota Masonic Cancer Center, Minneapolis, Minnesota, United States